CLINICAL TRIAL: NCT06792825
Title: HM2023-43: A Phase 2 Trial of Tafasitamab in Combination With Lenalidomide+Rituximab in Treatment-naive Follicular Lymphoma and Marginal Zone Lymphoma
Brief Title: HM2023-43:Ph 2 Trial of Tafasitamab With Lenalidomide+Rituximab in Treatment-naive FL and MZL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023LS183
Record Dates: First submitted 2025-01-23; First posted 2025-01-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — tafasitamab; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Follicular Lymphoma (Experimental): On Cycle 1, patients will receive an infusion of tafasitamab 12 mg/kg IV on Day 1, Day 8, Day 15 and day 22, rituximab 375 mg/m2 IV on Day 1, Day 8, Day 15 and Day 22, and lenalidomide 20 mg PO Day 1 through Day 21. On Cycles 2-3, patients will receive tafasitamab 12 mg/kg IV on Day 1, Day 8, Day 15 and day 22, rituximab 375 mg/m2 IV on day 1, and lenalidomide 20 mg PO Day 1-21. On Cycles 4-6, patients will receive an infusion of tafasitamab 12 mg/kg IV on Day 1, Rituximab 375 mg/m2 IV on Day 1, and lenalidomide 20 mg PO from Day 1-21. At the end of Cycle 6, patients on both cohorts will be assessed by Lugano standard. Patients in complete remission (CR) will continue on tafasitamab/rituximab and discontinue lenalidomide. Patients with partial response (PR) or stable disease (SD) will continue on all three drugs, tafasitamab/rituximab/lenalidomide, and if progressive disease (PD) will discontinue study.
  Interventions: Drug: Tafasitamab; Drug: Rituximab; Drug: Lenalidomide
- Marginal Zone Lymphoma (Experimental): On Cycle 1, patients will receive an infusion of tafasitamab 12 mg/kg IV on Day 1, Day 8, Day 15 and day 22, rituximab 375 mg/m2 IV on Day 1, Day 8, Day 15 and Day 22, and lenalidomide 20 mg PO Day 1 through Day 21. On Cycles 2-3, patients will receive tafasitamab 12 mg/kg IV on Day 1, Day 8, Day 15 and day 22, rituximab 375 mg/m2 IV on day 1, and lenalidomide 20 mg PO Day 1-21. On Cycles 4-6, patients will receive an infusion of tafasitamab 12 mg/kg IV on Day 1, Rituximab 375 mg/m2 IV on Day 1, and lenalidomide 20 mg PO from Day 1-21. At the end of Cycle 6, patients on both cohorts will be assessed by Lugano standard. Patients in complete remission (CR) will continue on tafasitamab/rituximab and discontinue lenalidomide. Patients with partial response (PR) or stable disease (SD) will continue on all three drugs, tafasitamab/rituximab/lenalidomide, and if progressive disease (PD) will discontinue study.
  Interventions: Drug: Tafasitamab; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Tafasitamab — Tafasitamab 12 mg/kg IV on Day 1, Day 8, Day 15 and day 22.
Drug: Rituximab — Rituximab 375 mg/m2 IV on day 1
  Other Names: R2
Drug: Lenalidomide — Lenalidomide 20 mg PO Day 1 through Day 21

SUMMARY:
The study follows a Simon's two-stage phase II trial design to evaluate the safety and efficacy of tafasitamab added to rituximab and lenalidomide for two treatment-naïve, parallel, independent cohorts: follicular lymphoma (FL) and marginal zone lymphoma (MZ). Each cohort, FL and MZ, will be evaluated separately. This study is presented to the patient and consent is signed prior to the initiation of treatment for their primary malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed marginal zone lymphoma
* Histologically confirmed CD20+ follicular lymphoma stage 1, 2 or 3a
* No prior systemic therapy for lymphoma
* Must be in need of treatment as evidenced by one or more of the following criteria:
* Bulky disease defined as:
* a nodal or extranodal (except spleen) mass >7cm in its greater diameter or,
* involvement of at least 3 nodal or extranodal sites (each with a diameter greater than >3 cm)
* Presence of at least one of the following B symptoms:
* fever (>38C) of unclear etiology
* night sweats
* weight loss greater than 10% within the prior 6 months
* Any other symptoms attributable to lymphomatous mass
* Endangerment of vital organ due to lymphomatous mass including but not limited to:
* Symptomatic or massive splenomegaly
* Compression syndrome (including but not limited to ureteral, orbital, gastrointestinal)
* Pleural, pericardial or ascitic effusion regardless of cell count
* Follicular lymphoma in leukemic phase (>5 X 109/L circulating cells)

OR:

* Follicular lymphoma graded high-risk by FLIPI2 score (see Appendix III)
* Adequate organ function within 14 days (28 days for pulmonary or cardiac) of study registration
* Participants who are of childbearing potential or have partners of child-bearing potential must agree to either total abstinence or use of both a highly effective (IUD, hormonal contraceptives, tubal ligation or vasectomy), and effective contraception (male or female condom, diaphragm or cervical cap) for the duration of treatment and for 12 months after the last dose of study drug.
* Able to tolerate prophylactic anticoagulation/antiplatelet therapy while on lenalidomide
* Able to provide written voluntary consent prior to the performance of any research related tests or procedures (or the subject's legally authorized representative (LAR) if enrollment of persons with diminished capacity is permitted - general permitted for Phase II and greater studies)

Exclusion Criteria:

* Seropositive for or active viral infection with hepatitis B virus (HBV):
* HBV surface antigen (HBsAg) positive
* HBV surface antigen (HBsAg) negative, HBV surface antibody (anti-HBs) positive and/or HBV core antibody (anti-HBc) positive, and detectable viral DNA
* Hepatitis C virus (HCV) positive subjects with chronic hepatitis C, or subjects with an active hepatitis C infection requiring anti-viral medication (at time of randomization).
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV).
* Prior history of lenalidomide use
* Prior history of malignancies, other than follicular or marginal zone lymphoma, unless the subject has been free of the disease for ≥ 5 years.
* Peripheral neuropathy ≥ grade 2 at time of screening
* Uncontrolled intercurrent illness.
* Active infection (requiring systemic therapy) or has received a live vaccine within 14 days prior to first dose of study drug.
* Presence or history of CNS involvement by lymphoma
* Patients who are not willing to take venous thromboembolic (VTE) prophylaxis or antiplatelet therapy
* Recent ( <1 year ) arterial thrombosis (any) or venous thrombosis ≥ grade 3 by CTCAE 5.0.
* Pregnant or breastfeeding as agents used in this study are Pregnancy Category X.

Women of childbearing potential must have two negative pregnancy tests (serum or urine) prior to their first dose of lenalidomide, and must agree to scheduled pregnancy testing while on treatment regardless of their birth control choice, per the requirements of the lenalidomide risk evaluation and mitigation strategy (REMS) program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2029-07-08 (Estimated); Study Completion 2031-07-08 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) | 1 year
  Estimate complete response (CR) at the end of study (after 12 cycles around 1 year) regimen of tafasitamab with lenalidomide and rituximab.

SECONDARY OUTCOMES:
Complete response (CR) | 6 months
  Estimate complete response (CR) rate after 6 cycles of treatment.
Overall response rate (ORR) | 1 year
  Estimate overall response rate (ORR) at the end of treatment (around 1 year).
Progression of disease (POD24) | 2 years
  Estimate progression of disease (POD24) within 24 months (2 years)
Progression free survival (PFS) | 3 years
  Estimate progression free survival (PFS) at 3 years after registration on study
Overall survival (OS) | 3 years
  Estimate overall survival (OS) at 3 years after registration on study
Rate of histologic conversion to DLBCL | 3 years
  Estimate rate of histologic conversion to DLBCL at any point on study.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided